CLINICAL TRIAL: NCT04309318
Title: Effects of Hemodynamic Changes Caused by Different Pneumoperitoneum Pressures on Cerebral Oxygenation in Laparoscopic Cholecystectomy
Brief Title: Effects of Hemodynamic Changes Caused by Different Pneumoperitoneum Pressure Ranges (10-12 mmHg and 13- 15 mmHg ) on Cerebral Oxygenation (With a Non-invasive Technique, Near Infrared Spectroscopy (NIRS) ) in Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, SEDAT SAYLAN, Assistant Professor, Karadeniz Technical University
Other Study IDs: 2020/11
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Pneumoperitoneum
Keywords: laparoscopic cholecystectomy; Pneumoperitoneum; Near Infrared Spectroscopy (NIRS)
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Low pneumoperitoneum (10-12 mmHg) pressure range group: Patients who have elective laparoscopic cholecystectomy with 10-12 mmHg intra-abdominal pneumoperitoneum pressure
  Interventions: Procedure: Low pneumoperitoneum (10-12 mmHg) pressure range group
- High pneumoperitoneum (13-15 mmHg) pressure range group: Patients who have elective laparoscopic cholecystectomy with 13-15 mmHg intra-abdominal pneumoperitoneum pressure
  Interventions: Procedure: High pneumoperitoneum (13-15 mmHg) pressure range group

INTERVENTIONS:
Procedure: Low pneumoperitoneum (10-12 mmHg) pressure range group — Patients who have elective laparoscopic surgery with 10-12 mmHg intra-abdominal pneumoperitoneum pressure
  Groups: Low pneumoperitoneum (10-12 mmHg) pressure range group
Procedure: High pneumoperitoneum (13-15 mmHg) pressure range group — Patients who have elective laparoscopic surgery with 13-15 mmHg intra-abdominal pneumoperitoneum pressure
  Groups: High pneumoperitoneum (13-15 mmHg) pressure range group

SUMMARY:
The negative effects of pneumoperitoneum used in laparoscopic cholecystectomy on cerebral metabolism, intracranial pressure, cardiovascular (blood pressure, heart rate, venous return) and respiratory system are known.

Pneumoperitoneum formed with low (10 - 12 mmHg) intraabdominal pressure causes less fluctuations in hemodynamic and respiratory changes. Previous studies have shown that intraabdominal pressure increase is effective on cerebral metabolism, leading to increased intracranial pressure.

The aim of this study is to investigate the hemodynamic effects of two different pneumoperitoneum pressure ranges (10-12 mmHg and 13-15 mmHg) on cerebral oxygenation with using Near Infrared Spectroscopy (NIRS), which is is a non-invasive technique, in laparoscopic cholecystectomy surgeries.

DETAILED DESCRIPTION:
The negative effects of pneumoperitoneum used in laparoscopic cholecystectomy on cerebral metabolism, intracranial pressure, cardiovascular (blood pressure, heart rate, venous return) and respiratory system are known.It is thought that pneumoperitoneum causes hemodynamic changes in the body by increasing blood catecholamine, vasopressin and norepinephrine levels.Sensitivity to these hemodynamic changes has been shown to be higher rate in patients with advanced age, morbid obesity, and increased intracranial pressure, and it is emphasized in studies that more attention should be paid to pneumoperitoneum pressures used in laparoscopic procedures with these groups.

In laparoscopic cholecystectomy surgery, pneumoperitoneum pressures used for surgical field visualization may differ.As a consequences, these different pressures have different haemodynamic and intracranial effects.Studies have shown that high intraabdominal pressure values cause more hemodynamic fluctuations than low intraabdominal pressure values.Systemic side effects have been shown to be lower in operations with low pneumoperitoneum pressure; In relation to the concept of multiple compartment syndrome, it is thought that the relationships between intraabdominal, intrathoracic and intracranial compartments, and changes in one compartment may affect other compartments and cause negative physiological and hemodynamic results.

There are studies in the literature on the hemodynamic effects of different pneumoperitoneum pressures.In our literature searches, we could not find any study comparing the effects of hemodynamic changes caused by two different pneumoperitoneum pressures, which can be classified as low and high, on cerebral oxygenation.We aimed to contribute to the literature by investigating the effects of different pneumoperitoneum pressure ranges on brain oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology (ASA) I-III,
* 18-65 years old
* under general anesthesia
* elective laparoscopic cholecystectomy

Exclusion Criteria:

* cerebrovascular diseases
* uncontrolled diabetes
* uncontrolled hypertension
* coagulopathy
* cirrhosis
* peritonitis
* asthma
* respiratory diseases such as chronic obstructive pulmonary disease (COPD)
* patients with morbid obesity
* multiple organ failure
* cases taken under emergency conditions
* cases returned to open cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic cholecystectomy between February 2020 and September 2020 at Karadeniz Technical University Faculty of Medicine Farabi Hospital under specified conditions
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Investigating the corelation between pneumoperitoneum pressure(mmHg) and brain oxygenation (with numeric NIRS value) | February 2020 - February 2021
  Investigating the effects of different pneumoperitoneum pressure ranges (10-12 mmHg and 13-15 mmHg) on brain oxygenation with NIRS (according to baseline NIRS value )

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No